CLINICAL TRIAL: NCT01496274
Title: A Phase II/III Open-label, Multicenter, Safety and Efficacy Study of a Recombinant Coagulation Factor IX Albumin Fusion Protein (rIX-FP) in Subjects With Hemophilia B
Brief Title: A Safety and Efficacy Study of a Recombinant Fusion Protein Linking Coagulation Factor IX With Albumin (rIX-FP) in Patients With Hemophilia B
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSL654_3001; 2011-002415-28 (EudraCT Number)
Record Dates: First submitted 2011-12-19; First posted 2011-12-21 (Estimated); Results first posted 2016-05-09 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-04

CONDITIONS: Hemophilia B
MeSH Terms: conditions — Hemophilia B | interventions — albutrepenonacog alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prophylaxis (Experimental): Routine weekly prophylaxis and episodic treatment for bleeding episodes. An individualized dosing interval may be tested in sub-group subjects during the 2nd part of the trial.
  Subjects may participate in a surgical 'sub-study' in which rIX-FP may be administered prior to, during and after surgical intervention.
  Interventions: Biological: rIX-FP
- On-demand (Experimental): Episodic treatment for bleeding episodes during the first 6 months then switch to routine weekly prophylaxis for a further 6 months Subjects may participate in a surgical 'sub-study' in which rIX-FP may be administered prior to, during and after surgical intervention.
  Interventions: Biological: rIX-FP

INTERVENTIONS:
Biological: rIX-FP — Recombinant IX-FP (rIX-FP) is a fusion protein linking coagulation factor IX with albumin, and will be administered by intravenous administration

SUMMARY:
This study will examine the safety, pharmacokinetics and efficacy of rIX-FP for the control and prevention of bleeding episodes in subjects who have previously received factor replacement therapy for hemophilia B.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects, 12 to 65 years old
* Severe hemophilia B (FIX activity of ≤ 2%)
* Subjects who have received FIX products (plasma-derived and/or recombinant FIX) for > 150 exposure days (EDs)
* No history of FIX inhibitor formation, no detectable inhibitors at Screening and no family history of inhibitors against FIX
* Written informed consent for study participation
* On-demand subjects only, who have experienced a minimum average of 2 non-trauma induced bleeding episodes requiring treatment with a FIX product during the previous 6 or 3 months

Exclusion Criteria:

* Known hypersensitivity to any FIX product or hamster protein
* Known congenital or acquired coagulation disorder other than congenital FIX deficiency
* HIV positive subjects with a CD4 count < 200/mm3
* Low platelet count, kidney or liver dysfunction
* Recent life-threatening bleeding episode

Ages: 12 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2012-02; Primary Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Program Director, Study Director — CSL Behring
Locations (30):
- United States (4):
  - Rush University Medical Center, Chicago, Illinois
  - Indiana Hemophilia and Thrombosis Center, Inc., Indianapolis, Indiana
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - BloodCenter of Wisconsin, Milwaukee, Wisconsin
- AKH Wien [Hämatologie, Hämostaseol, Vienna, Austria
- SHAT "Joan Pavel" OOD [Hemorrhagic Diathesis and Anemia], Sofia, Bulgaria
- France (4):
  - Centre Hospitalier Universitaire de Brest/CHU Morvan, Brest
  - C.R.T.H. Hôp. Bicêtre-Hémophilie, Le Kremlin-Bicêtre
  - CHU de Lyon - Hôpital Edouard Herriot [Hemophilie], Lyon
  - Hôpital Necker-CRTH, Paris
- Germany (5):
  - Instit. für Experimentelle - Hämato & Transfusionsmedizin, Bonn
  - Zentralkrankenhaus Prof. Hess-Kinderklinik, Bremen
  - Unikinderklinik Frankfurt/Main [Kinderheilkunde], Frankfurt
  - Universitätsklinikum Hamburg-Eppendorf, Abt für Pädiatr. Hämatologie, Hamburg
  - Werlhof-Inst. Hannover, Hanover
- Chaim Sheba Medical Center, Tel Aviv, Israel
- Italy (3):
  - IRCCS Ospedale Maggiore[Centro emofilia e Trombosi], Milan
  - A.O.U. di Parma [Centro di Rif. Reg. per la cura dell'Emofil, Parma
  - Osp. S.Bortolo ULSS N.6 [Terapie Cell. ed Ematologia], Vicenza
- Japan (7):
  - Nara Medical University Hospital [PEDIATRICS], Kashihara
  - University of Occupational and Environmental Health, Kitakyushu
  - Nagoya University Hospital, Nagoya
  - The Hospital of Hyogo College of Medicine, Nishinomiya
  - Ogikubo Hospital, Tokyo
  - Tokyo Medical University Hospital, Tokyo
  - St. Marianna University, School of Medicine, Yokohama Seibu, Yokohama
- FGU "Kirov Research Institute of Haemotology and Blood Trans, Kirov, Russia
- Spain (3):
  - C.H.U. A Coruña [Hematología], A Coruña
  - H.U.Vall d'Hebrón [Hemofillia], Barcelona
  - H.U. La Paz [Coagulopatias Congénitas], Madrid

REFERENCES:
- [Derived] Santagostino E, Martinowitz U, Lissitchkov T, Pan-Petesch B, Hanabusa H, Oldenburg J, Boggio L, Negrier C, Pabinger I, von Depka Prondzinski M, Altisent C, Castaman G, Yamamoto K, Alvarez-Roman MT, Voigt C, Blackman N, Jacobs I; PROLONG-9FP Investigators Study Group. Long-acting recombinant coagulation factor IX albumin fusion protein (rIX-FP) in hemophilia B: results of a phase 3 trial. Blood. 2016 Apr 7;127(14):1761-9. doi: 10.1182/blood-2015-09-669234. Epub 2016 Jan 11. PMID 26755710

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 30 sites in 10 countries.
Pre-assignment Details: A total of 69 subjects provided informed consent and were screened for study participation. Of these, 63 subjects were enrolled and treated with rIX-FP.
Groups:
- On-demand: Episodic treatment for bleeding episodes for up to 26 weeks then switch to routine weekly prophylaxis for the remainder of the study.
  Subjects may participate in a surgical 'sub-study' in which rIX-FP may be administered prior to, during and after surgical intervention.
Period: Overall Study
Arm/Group | Prophylaxis | On-demand
Started | 40 | 23
Completed | 37 | 18
Not Completed | 3 | 5
Not completed — Protocol Violation | 0 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 0 | 3

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Prophylaxis: Routine weekly prophylaxis and episodic treatment for bleeding episodes. An individualized dosing interval may be tested in sub-group subjects during the 2nd part of the trial.
  Subjects may participate in a surgical 'sub-study' in which rIX-FP may be administered prior to, during and after surgical intervention.
  rIX-FP: Recombinant IX-FP (rIX-FP) is a fusion protein linking coagulation factor IX with albumin, and will be administered by intravenous administration
- On-demand: Episodic treatment for bleeding episodes for up to 26 weeks then switch to routine weekly prophylaxis for the remainder of the study.
  Subjects may participate in a surgical 'sub-study' in which rIX-FP may be administered prior to, during and after surgical intervention.
  rIX-FP: Recombinant IX-FP (rIX-FP) is a fusion protein linking coagulation factor IX with albumin, and will be administered by intravenous administration
- Total: Total of all reporting groups
Arm/Group | Prophylaxis | On-demand | Total
Number analyzed (Participants) | 40 | 23 | 63
Age, Customized [Number; unit: participants]
  0 to 11 years | 0 | 0 | 0
  12 to 17 years | 7 | 0 | 7
  18 to 64 years | 33 | 23 | 56
  65 years and over | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 40 | 23 | 63

OUTCOME MEASURES:

1. Primary Outcome: Change in Frequency of Spontaneous Bleeding Events Between On-demand and Prophylaxis Treatments (Annualized)
Description: Subjects in the on-demand arm received on-demand dosing with rIX-FP for up to 26 weeks (on-demand regimen), and then received weekly prophylaxis with rIX-FP for the remainder of the study (prophylaxis regimen). The effectiveness of prophylaxis in comparison to on-demand therapy was investigated by comparing the same subject's annualized spontaneous bleeding rate (AsBR) during the on-demand regimen and during the prophylaxis regimen.
Time Frame: Up to 26 weeks for on-demand regimen, and between 1 and 17 months for prophylaxis regimen.
Population: This analysis includes only the participants assigned to the on-demand arm who received at least 1 dose of rIX-FP in the on-demand regimen and at least 1 dose of rIX-FP in the prophylaxis regimen.
Measure: Median (Inter-Quartile Range); unit: bleeds/year/subject
Groups:
- On-demand Arm, On-demand Regimen: Participants in the On-demand Arm, when receiving episodic treatment for bleeding episodes (on-demand regimen).
- On-demand Arm, Prophylaxis Regimen: Participants in the On-demand Arm, when receiving routine weekly prophylaxis (prophylaxis regimen).
Arm/Group | On-demand Arm, On-demand Regimen | On-demand Arm, Prophylaxis Regimen
Number analyzed (Participants) | 19 | 19
bleeds/year/subject | 15.43 [7.98 to 17.96] | 0.00 [0.00 to 0.96]
Statistical Analysis 1: Comparison: On-demand Arm, On-demand Regimen vs On-demand Arm, Prophylaxis Regimen; A test of null hypothesis that the ratio of AsBR (prophylaxis regimen/on-demand regimen) was ≥ 0.50 was conducted at the 1-sided 0.025 level. Matched pairs design with 19 subjects and 2 observations per subject; Test type: Superiority or Other; p < 0.0001, Wilcoxon signed-rank test — P value is based on a Wilcoxon signed-rank test of H0: AsBR ratio (prophylaxis regimen/on-demand regimen) ≥ 0.50. The ratio was based on the original scale

2. Primary Outcome: Number of Subjects Developing Inhibitors Against Factor IX (FIX)
Description: The number of participants developing inhibitors against factor IX (FIX) along with the 95% Clopper-Pearson confidence interval, are summarized for subjects with 50 or more exposure days (EDs) to rIX-FP, and for all participants in the study.
Time Frame: Up to 27.7 months (maximum)
Population: Safety Population
Measure: Number (95% Confidence Interval); unit: participants
Groups:
- Safety Population: The Safety population consisted of subjects who received at least 1 dose of rIX-FP during the study.
Arm/Group | Safety Population
Number analyzed (Participants) | 63
participants
  Participants with >=50 EDs to rIX-FP (n = 49) | 0 [0.0 to 7.3]
  All participants (n = 63) | 0 [0.0 to 5.7]

3. Secondary Outcome: The Frequency of Related Adverse Events
Description: The percentage of participants experiencing treatment-related adverse-events (TEAEs).
Time Frame: For the duration of the study; median 20.27 months.
Population: Safety Population
Measure: Number; unit: Percentage of participants
Arm/Group | Prophylaxis | On-demand | Safety Population
Number analyzed (Participants) | 40 | 23 | 63
Percentage of participants
  Related TEAE | 10.0 | 4.3 | 7.9
  Not related TEAE | 87.5 | 78.3 | 84.1

4. Secondary Outcome: Number of Subjects Developing Antibodies Against rIX-FP
Time Frame: For the duration of the study; median 20.27 months.
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Safety Population
Number analyzed (Participants) | 63
participants | 0

5. Secondary Outcome: Proportion of Bleeding Episodes Requiring One or ≤ Two Injections of rIX-FP to Achieve Hemostasis
Description: Number of injections required to achieve hemostasis expressed as a percentage of the bleeding episodes requiring treatment.
Time Frame: For the duration of the study; median 20.27 months.
Population: Efficacy Population
Measure: Number; unit: percentage of bleeding episodes treated
Units Other Than Participants: bleeding episodes requiring treatment
Arm/Group | Prophylaxis | On-demand Arm, On-demand Regimen | On-demand Arm, Prophylaxis Regimen
Number analyzed (Participants) | 40 | 23 | 19
Number analyzed (bleeding episodes requiring treatment) | 101 | 220 | 37
percentage of bleeding episodes treated
  1 injection | 92.1 | 94.5 | 91.9
  1 or 2 injections | 100.0 | 98.6 | 94.6

6. Secondary Outcome: Investigator's Overall Clinical Assessment of Hemostatic Efficacy for Treatment of Bleeding Episodes, Based on a Four Point Ordinal Scales (Excellent, Good, Moderate, Poor/No Response)
Description: Number of bleeding episodes requiring treatment that resulted in hemostatic efficacy of excellent, good, moderate, poor/no response, according to the Investigator's clinical assessment of hemostatic efficacy, expressed as a percentage of the bleeding episodes requiring treatment.
Time Frame: For the duration of the study; median 20.27 months
Population: Efficacy Population
Measure: Number; unit: percentage of bleeding episodes
Units Other Than Participants: bleeding episodes requiring treatment
Arm/Group | Prophylaxis | On-demand
Number analyzed (Participants) | 40 | 23
Number analyzed (bleeding episodes requiring treatment) | 101 | 257
percentage of bleeding episodes
  Excellent | 71.3 | 87.5
  Good | 20.8 | 7.4
  Moderate | 3.0 | 2.3
  Poor/No response | 0 | 0.4
  Missing | 5.0 | 2.3

7. Secondary Outcome: rIX-FP Consumed Per Month While Maintaining Assigned Prophylactic Treatment Interval During Routine Prophylaxis.
Description: Time frame: For Prophylaxis Arm 7-, 10- and 14-day regimens, median 269, 240 and 386 days respectively. For On-demand Arm, prophylaxis regimen, median 316 days.
Time Frame: Median 269, 240, 386 and 316 days, respectively (see Description)
Population: Efficacy Population
Measure: Mean (Standard Deviation); unit: IU/kg/month
Groups:
- Prophylaxis Arm, 7-day Regimen: Subjects received prophylactic rIX-FP on a weekly basis.
- Prophylaxis Arm, 10-day Regimen: Subjects received prophylactic rIX-FP every 10 days.
- Prophylaxis Arm, 14-day Regimen: Subjects received prophylactic rIX-FP every 14 days.
Arm/Group | On-demand Arm, Prophylaxis Regimen | Prophylaxis Arm, 7-day Regimen | Prophylaxis Arm, 10-day Regimen | Prophylaxis Arm, 14-day Regimen
Number analyzed (Participants) | 19 | 40 | 7 | 21
IU/kg/month | 191.69 (36.33) | 202.68 (47.92) | 201.50 (42.56) | 157.44 (16.34)

8. Secondary Outcome: Incremental Recovery of rIX-FP
Description: Pharmacokinetic (PK) data are presented for a single 50 IU/kg dose of rIX-FP.
Time Frame: 336 hours
Population: The PK population comprised 46 subjects who received at least 1 dose of rIX-FP at 50 IU/kg. Data are presented for subjects from the PK population who had a sufficient number of analyzable PK samples for evaluation of the PK profile of rIX-FP.
Measure: Mean (Standard Deviation); unit: (IU/dL)/(IU/kg)
Arm/Group | Prophylaxis | On-demand
Number analyzed (Participants) | 27 | 18
(IU/dL)/(IU/kg) | 1.29 (0.33) | 1.24 (0.25)

9. Secondary Outcome: Half-life (t1/2) of a Single Dose of rIX-FP
Description: PK data are presented for a single 50 IU/kg dose of rIX-FP.
Time Frame: 336 hours
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hour
Groups:
- On-demand: Episodic treatment for bleeding episodes up to 26 weeks then switch to routine weekly prophylaxis for the remainder of the study.
  Subjects may participate in a surgical 'sub-study' in which rIX-FP may be administered prior to, during and after surgical intervention.
Arm/Group | Prophylaxis | On-demand
Number analyzed (Participants) | 26 | 17
hour | 104.77 (22.73) | 96.88 (20.94)

10. Secondary Outcome: Area Under the Curve (AUC)
Description: AUC to the last sample with quantifiable drug concentration (AUClast) of a single dose of rIX-FP. PK data are presented for a single 50 IU/kg dose of rIX-FP.
Time Frame: 336 hours
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: IU*hr/dL
Arm/Group | Prophylaxis | On-demand
Number analyzed (Participants) | 27 | 18
IU*hr/dL | 6534.15 (1856.96) | 5963.30 (1893.00)

11. Secondary Outcome: Clearance of a Single Dose of rIX-FP
Description: PK data are presented for a single 50 IU/kg dose of rIX-FP.
Time Frame: 336 hours
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mL/hr
Arm/Group | Prophylaxis | On-demand
Number analyzed (Participants) | 26 | 17
mL/hr | 50.19 (12.92) | 59.00 (19.37)

12. Secondary Outcome: Investigator's (or Surgeon's) Overall Clinical Assessment of Hemostatic Efficacy for Surgical Prophylaxis, Based on a Four Point Ordinal Scale (Excellent, Good, Moderate, Poor/No Response)
Description: Number of surgical events treated prophylactically with rIX-FP that resulted in hemostatic efficacy of excellent, good, moderate, poor/no response, according to the Investigator's (surgeon's) overall assessment of hemostatic efficacy for surgical prophylaxis.
Time Frame: Up to 14 days after surgery
Population: Surgical Population
Measure: Number; unit: events
Units Other Than Participants: events
Groups:
- Surgical Population: The Surgical population consisted of 3 subjects in the prophylaxis arm and 1 subject in the on demand arm who received at least 1 dose of rIX FP for a major or minor surgical procedure.
Arm/Group | Surgical Population
Number analyzed (Participants) | 4
Number analyzed (events) | 6
events
  Excellent | 6
  Good | 0
  Moderate | 0
  Poor/No response | 0

13. Secondary Outcome: Annualized Spontaneous Bleeding Events Compared Between 7 Day Prophylactic and Extended Regimens
Description: Median number of spontaneous bleeds per year per subject comparing 7-, 10- and 14- day prophylactic regimens.
Time Frame: During treatment, between median 240 and 386 days per subject.
Population: Efficacy Population
Measure: Median (Inter-Quartile Range); unit: bleeds/year/subject
Arm/Group | Prophylaxis Arm, 7-day Regimen | Prophylaxis Arm, 10-day Regimen | Prophylaxis Arm, 14-day Regimen
Number analyzed (Participants) | 38 | 7 | 21
bleeds/year/subject | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 1.00]

ADVERSE EVENTS:
Time Frame: For the duration of the study, up to 27.7 months.
Description: The Safety analysis population consisted of subjects who received at least 1 dose of rIX-FP during the study. Adverse Event (AE) data are treatment-emergent data unless otherwise noted.
  The total number of participants in the number affected by Other (non-serious) AEs, is the total number of participants experiencing at least one non-serious AE.
Arm/Group | Prophylaxis | On-demand
Serious Adverse Events (participants affected / at risk) | 1/40 | 2/23
Other Adverse Events (participants affected / at risk) | 36/40 | 18/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prophylaxis (N=40) | On-demand (N=23)
ACQUIRED EPILEPTIC APHASIA (Nervous system disorders) | 0 (0) | 1 (1)
SYNOVITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — This serious adverse event was not treatment-emergent.
MUSCLE HAEMORRHAGE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — This serious adverse event was not treatment-emergent.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prophylaxis (N=40) | On-demand (N=23)
LIMB INJURY (Injury, poisoning and procedural complications) | 5 (5) | 1 (1)
CONTUSION (Injury, poisoning and procedural complications) | 3 (5) | 1 (3)
LACERATION (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
HEADACHE (Nervous system disorders) | 11 (26) | 4 (8)
DIZZINESS (Nervous system disorders) | 4 (5) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 2 (2) | 3 (4)
TOOTHACHE (Gastrointestinal disorders) | 4 (4) | 1 (1)
ACNE (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 9 (19) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (3)
SYNOVITIS (Musculoskeletal and connective tissue disorders) | 3 (6) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
TENDONITIS (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 10 (27) | 6 (11)
INFLUENZA (Infections and infestations) | 4 (7) | 3 (3)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 5 (7) | 0 (0)
BRONCHITIS (Infections and infestations) | 4 (4) | 1 (1)
PHARYNGITIS (Infections and infestations) | 3 (3) | 2 (2)
GASTROENTERITIS (Infections and infestations) | 3 (4) | 0 (0)
ACUTE TONSILLITIS (Infections and infestations) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
CSL agreements and restrictions on publishing may vary with individual investigators; however, CSL will not prohibit any investigator from publishing. CSL supports the publication of results from all centers of a multi-center trial and generally requires that reports based on single-site data not precede the primary publication of the entire clinical trial.